CLINICAL TRIAL: NCT04967339
Title: A Randomized Control Trial in Patients With Medial Knee Osteoarthritis Comparing the Clinical and Biomechanical Effect of Foot Deformity Correcting Insoles and Lateral Wedge Insoles
Brief Title: Comparison of Different Insoles as Conservative Treatment for Medial Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-InsoleStudy
Record Dates: First submitted 2021-07-13; First posted 2021-07-19 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Osteoarthritis, Knee
Keywords: Mediale Knee Osteoarthritis; Conservative Treatment; Insoles
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Foot deformity correcting insole arm (Experimental): Patients allocated to the "foot deformity correcting insole" arm will receive insoles to correct their foot deformities (plano-valgus foot deformity).
  Interventions: Device: Foot deformity correcting insoles
- Lateral wedge insole arm (Active Comparator): Patient allocated to the "Lateral wedge insole" arm will receive conventional lateral wedge insole.
  Interventions: Device: Lateral wedge insoles

INTERVENTIONS:
Device: Foot deformity correcting insoles — Foot deformity correcting insoles (e.g. insoles with medial arch support for plano-valgus deformity)
  Arms: Foot deformity correcting insole arm
Device: Lateral wedge insoles — Lateral wedge insoles
  Arms: Lateral wedge insole arm

SUMMARY:
In patients with early to mid-stage knee osteoarthritis (OA), a conservative treatment is indicated. In medial knee OA (when mainly the medial compartment of the knee is affected by OA), lateral wedge insoles have been promoted as cost effective and simple solution. However, clinical trials report conflicting results, with some reporting no benefit while others reported a small decrease in knee pain. Recent studies reported medial OA patients to have a tendency to a plano-valgus foot deformity, which is associated with a varus lower limb alignment and an internal rotation of the tibia. Some authors thus proposed the correction of plano-valgus deformity with foot deformity correcting insoles instead of lateral wedge insoles. Until today, only one study investigated the effect of foot deformity correcting insoles (e.g. with medial arch support) as alternative to lateral wedge insoles and reported encouraging results. However, they used lateral wedge insoles with custom arch support instead of foot deformity correcting customized insoles along (without lateral wedge). Furthermore, they did not perform any biomechanical analyses. The primary object of this study is to compare the effect of foot deformity correcting insoles for plano-valgus foot deformities and lateral wedge insoles on knee load distribution, knee pain and patient reported outcome measures in early to mid-stage medial knee OA patients after 6 and 12 months.

DETAILED DESCRIPTION:
Osteoarthritis (OA) of the knee is defined as an inflammatory process leading to loss of protective cartilage which results in pain, disability and loss of function. Around 25% of the population between 55 and 84 years is affected by OA of the knee. It can be graded using various classification, one of the most used being the Kellgren-Lawrence-Score (KL) ranging from 1 (early) to 4 (end stage). The treatment of choice for end-stage three compartmental knee OA (KL 4) is a total knee arthroplasty (TKA), whereby the damaged/degenerated parts of the knee are removed and replaced by a prosthesis. However, in patients with early to mid-stage OA (KL 1-3), which are usually younger patients, a conservative treatment is indicated. The goal of this conservative treatment is to relieve symptoms and at best slow progression of the diseases.

In medial knee OA (when mainly the medial compartment of the knee is affected by OA), one approach is to reduce the medial compartment contact force (MCF) by shifting load from the medial (disease affected) to lateral (disease free) compartment. Thereby lateral wedge insoles have been promoted as cost effective and simple solution. The biomechanical idea of these insoles is a shift in load distribution through a change in lower limb alignment. The lateral wedge of the insoles leads to a change in foot alignment (varus hindfoot) and consequently to a change in knee alignment (valgus knee = "knock-knees") and load distribution. Biomechanical studies confirmed a reduction in external knee adduction moment (EKAM) and knee adduction angular impulse (KAAI), which are surrogate measures to estimate knee joint load distribution (e.g. MCF). However, clinical trials report conflicting results, with some reporting no benefit while others reported a small decrease in knee pain in at least some patients.

In the light of this, the connection between knee OA and foot deformities has been reassessed. One study found patients with medial knee OA to have a more pronated foot type (i.e. tendency to plano-valgus deformity) compared to an age-matched control group without OA. Other investigations found more rigid foot types in patients with medial knee OA and a more internally rotated tibia during gait as well as an inversion of the forefoot. This seems important because the hindfoot axis has a significant influence on the mechanical axis of the lower limb and thereby on the load distribution in the knee. Half a degree valgisation of the hindfoot axis leads to one-degree varisation of the mechanical axis. Furthermore, a plano-valgus foot morphology was found to lead to internal rotation of the tibia which increases shear forces in the medial knee compartment.

In summary, patients with medial knee OA tend to have a plano-valgus foot deformity which is associated with a varus lower limb alignment and an internal rotation of the tibia. Both have been associated to an increased loading of the medial compartment. Consequently, some authors proposed the correction of plano-valgus deformity with customized foot deformity correcting insoles instead of lateral wedge insoles as conservative treatment option for early to mid-stage medial knee OA. Until today, only one study investigated the effect of foot deformity correcting insoles (e.g. insoles with customized medial arch support) as alternative to lateral wedge insoles and reported encouraging results. However, they used lateral wedge insoles with and without medial arch support and did not explicitly only correct the foot deformity. Furthermore, they did not perform any biomechanical analysis, which seems important since some previous studies found significant differences in KAAI and EKAM among patients.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* Aged between 40 to 80 years
* Early to mid-stage (KL 1 - 3) OA of the medial compartment of the knee based on X-ray and MRI images
* Plano-valgus foot deformity based on clinical assessment
* Availability of conventional radiographs, long-leg films, and a knee-MRI no older than 1 year at time of inclusion
* Ability to walk without walking aid for more than 15min

Exclusion Criteria:

* Contraindications and limitations of the MD as described in the instructions for use.
* Inability to follow the procedures of the investigation, e.g. due to language problems, psychological disorders, dementia, etc. of the subject,
* Enrolment of the PI, his/her family members, employees and other dependent persons
* Relevant OA (Kellgren-Lawrence-Score >2) of the lateral compartment of the knee based on X-ray and MRI images
* BMI higher than 40 kg/m
* Fix varus deformities over 20 degrees
* Neurological or rheumatoid diseases of any kind
* History of high tibial osteotomy, other realignment surgery of the knee or foot
* Foot or ankle problems that contraindicated the use of footwear load-modifying interventions
* Relevant ligamentous instability

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Numeric pain scale (NRS) | pre-treatment
Numeric pain scale (NRS) | 3 months
Numeric pain scale (NRS) | 6 months
Numeric pain scale (NRS) | 12 months
External knee adduction moment (EKAM) | pre-treatment
External knee adduction moment (EKAM) | 3 months
External knee adduction moment (EKAM) | 6 months
External knee adduction moment (EKAM) | 12 months
Knee adduction angular impulse (KAAI) | pre-treatment
Knee adduction angular impulse (KAAI) | 3 months
Knee adduction angular impulse (KAAI) | 6 months
Knee adduction angular impulse (KAAI) | 12 months
Western Ontario and McMaster OA Index (WOMAC) | pre-treatment
Western Ontario and McMaster OA Index (WOMAC) | 3 months
Western Ontario and McMaster OA Index (WOMAC) | 6 months
Western Ontario and McMaster OA Index (WOMAC) | 9 months
Western Ontario and McMaster OA Index (WOMAC) | 12 months
Knee Injury and Osteoarthritis Outcome Score (KOOS) | pre-treatment
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 3 months
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 6 months
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 12 months
Oxford-12 Knee Score (OKS) | pre-treatment
Oxford-12 Knee Score (OKS) | 3 months
Oxford-12 Knee Score (OKS) | 6 months
Oxford-12 Knee Score (OKS) | 12 months
Knee Society Score (KSS) | pre-treatment
Knee Society Score (KSS) | 3 months
Knee Society Score (KSS) | 6 months
Knee Society Score (KSS) | 12 months
EQ-5D | pre-treatment
EQ-5D | 3 months
EQ-5D | 6 months
EQ-5D | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Frank Klenke, Prof, Principal Investigator — Universitätsklinik für Orthopädische Chirurgie und Traumatologie Inselspital
Locations (1):
- Universitätsklinik für Orthopädische Chirurgie und Traumatologie Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No